CLINICAL TRIAL: NCT04011319
Title: Group Culture May Affect Human Embryo Quality in Assisted Reproduction Technology
Brief Title: Group Culture May Affect Embryo Quality in Assisted Reproduction Technology
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Tang-Du Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCIEQ
Record Dates: First submitted 2019-03-31; First posted 2019-07-08 (Actual); Last update posted 2019-07-08 (Actual); Status verified 2019-06

CONDITIONS: Embryo Quality
Keywords: Group culture; Embryo quality; Implantation rate; Clinical pregnancy

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- convention culture (No Intervention): Each droplet separate culturing an individual embryo.
- group culture (Experimental): Embryos were cultured in the same droplet.
  Interventions: Behavioral: group culture

INTERVENTIONS:
Behavioral: group culture — Four embryos were cultured in the same droplet by a special dish.
  Arms: group culture

SUMMARY:
One of the vital factors in achieving pregnancies in assisted reproductive technologies (ART) is maximizing embryo quality, which is significantly influenced by embryo culture conditions. A microwell culture system that facilitates group culture, improves embryonic development. The investigators use a new special culture dish to examine the effect of group culture on embryonic development in vitro. Zygotes derived from sibling oocytes were completely denuded from cumulus cells and spermatozoa, then randomly divided into conventional droplet culture or group culture. Embryos cultured in microwell system (group culture) were compared to conventional droplet culture (one zygote per drop). Relevant parameters are recorded to evaluate the validity of group culture in ART.

DETAILED DESCRIPTION:
Providing optimal culture conditions for the embryos in ART is crucial, due to its high impact on embryo development and thus on the pregnancy outcome. Several strategies have been proposed in order to improve embryo culture conditions and clinical pregnancy rates. Currently, the establishment of autocrine and paracrine communications and embryo-to-embryo interactions should contribute to the detoxification of the culture medium, facilitating embryo development and improving the implantation rate. Many studies have provided evidence related to the impact of group culture condition on the success of the embryonic development in animals. But the advantage of group culture to improve the embryonic development and pregnancy outcomes of ART in human remains elusive. Therefore, the investigator aim to discuss the effectiveness of group culture in ART.

In this study, zygotes derived from sibling oocytes were randomized 1:1 to either the microwell group culture (experiment group) or conventional droplet culture (control group). In experiment group, 4 zygotes cultured in a new special microwell (120 μl droplet were divided into 4 areas) with a corral dish (EMBC-010, LifeGlobal), embryos can communicate with each other in the same culture environment. In control group, single embryo individually cultured in a droplet (60 μl). Embryos were cultured in specific desktop three-gas incubators (COOK) of 37°C, 6% CO2 (carbon dioxide) , 5% O2 and 89% N2, and scored according to the criteria described in the ESHRE-ALPHA consensus. Consequently, exploitable embryos rate, good embryo quality, blastocyst formation rate were recorded. Other relevant parameters such as clinical pregnancy, live-birth or miscarriage were also recorded to evaluate the outcomes. Proper culture conditions can result in superior embryo viability, this research intends to discuss whether group culture can improve the embryo quality and clinical outcomes in ART.

ELIGIBILITY:
Inclusion Criteria:

* Patients undergoing IVF/ICSI cycle.
* Number of oocytes≥ 8.

Exclusion Criteria:

* Number of mature oocytes less than 6.
* The number of normal fertilized zygotes less than 4.

Ages: 22 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 2000 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
Efficacy of group culture on embryo potential | 1 year
  Embryo potential was evaluated by the clinical pregnancy rate

CONTACTS AND LOCATIONS:
Overall Officials: Bo Li, Study Director — Tang-Du Hospital
Locations (1):
- Tangdu Hospital, Xi'an, Shaanxi, China